CLINICAL TRIAL: NCT03629301
Title: Efficacy of an Internet-delivered Intervention Based on the Diabetes Prevention Program for Weight Loss in Overweight and Obese Mexican Adults: 3 and 6 Months Randomized Controlled Trial
Brief Title: Obesity Treatment Using an Internet-delivered Intervention Based on the Diabetes Prevention Program in Mexican Adults
Acronym: DPPON-MEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Sonora (Other)
Responsible Party: Principal Investigator, Rolando Giovanni Díaz Zavala, Principal Investigator, Universidad de Sonora
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USO313003634
Record Dates: First submitted 2018-08-10; First posted 2018-08-14 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Obesity or Overweight
Keywords: Obesity; Overweight; Lifestyle Intervention; Randomized controlled Trial; Internet delivered; Online; Weight loss
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ID-DPP group (Experimental): Internet-delivered intervention based on the DPP
  Interventions: Behavioral: ID-DPP group
- Wait-list Group (Other)
  Interventions: Other: Wait-list Group

INTERVENTIONS:
Behavioral: ID-DPP group — This group will receive a 6 month long online behavioral change protocol adapted from the Diabetes Prevention Program. It includes 18 sessions, 12 delivered weekly (during the first 3 months) and 6 delivered biweekly (during the last 3 month period). A web page will be used to deliver the sessions, while the nutritional counseling will be delivered using video calls via Facebook chat. Participants will receive an hypocaloric (1200-1800 kcal, carbohydrates: 45-65%, fats: 20-35% and protein: 10-35%), personalized diet.
  Arms: ID-DPP group
Other: Wait-list Group — This group will only receive written information with recommendations on healthy eating. When the study has finished this group will receive a behavioral change protocol with nutritional counseling using a face-to-face format.
  Arms: Wait-list Group

SUMMARY:
In Mexico, 7 out of 10 adults are overweight or obese. The diseases associated with these conditions (diabetes, cardiovascular disease and some cancers) are those that impact the most on the disability-adjusted life years of Mexicans and on their mortality rates. A reduction in body weight of 5-10% can reduce the incidence of obesity related diseases. The gold standard for treating obesity is an intensive lifestyle change program such as the Diabetes Prevention Program (DPP) whose effectiveness has been evaluated in various formats and populations with positive results, including in Mexico. However, the DPP is not accessible to all sectors of the population. To increase its dissemination, the implementation of online interventions based on the DPP (oi-DPP) has been proposed. A systematic review of oi-DPP showed promising results, however, the evidence is limited and the lack of studies of high methodological quality is highlighted. The main objective of this project is to evaluate the efficacy of an oi-DPP for weight loss in Mexican adults with overweight or obesity at 3 months. The study design is a randomized controlled trial with 2 arms: oi-DPP and wait-list control. A 3 months pilot study (n=30) will be conducted prior to the main study to estimate sample size, considering an alpha error of 0.05 and power of 80%. The primary outcome is the mean change in body weight from baseline to 3 months post-baseline between the 2 groups. Secondarily, differences in biochemical parameters (fasting glucose, total cholesterol, LDL cholesterol, HDL cholesterol, triglycerides and gamma glutamyl transferase) from baseline to 3 months will be evaluated, as well as mean changes from baseline to 3 and 6 months in body mass index, waist circumference, systolic and diastolic blood pressure, depression and quality of life scales and the number of participants achieving a weight loss greater than 5% of initial body weight. Body weight will be also evaluated at 6 months post-baseline. The previous measurements will apply both in the pilot study and the study except for the biochemical parameters that will only be included in the main study. The differences between the 2 groups for each variable will be analyzed using a t test for independent samples, in case of having a parametric sample. Otherwise, the Mann-Whitney U test will be used. Analysis will follow the intent-to-treat principle.

ELIGIBILITY:
Inclusion Criteria:

* Mexican adults (≥ 18 years and ≤60)
* Residents of the city of Hermosillo, Sonora
* Overweight or obese (BMI ≥ 25 and ≤45)
* Internet access at home
* Basic computer skills
* Facebook active account
* Candidates must make records of their food consumption for 5 days.

Exclusion Criteria:

* Substance abuse
* Consumption of more than 14 alcoholic beverages per week (equivalent to 280 g of alcohol)
* Diagnosis of psychiatric conditions that could prevent adherence to treatment
* Previous diagnosis of medical conditions with significant effect on body weight
* Diagnosis of diabetes
* Systolic blood pressure> 160 mm / Hg
* Pregnant women who are breastfeeding or who plan to become pregnant during the study period
* Consumption of medications with an effect on body weight such as metformin, orlistat or glucocorticoids.
* Participating in another program to reduce weight or performing structured physical exercise other than walking> 180 min / week
* Plan to participate in some treatment for weight loss during the study
* Any other condition in which weight loss or physical activity is contraindicated
* Previous diagnosis of kidney failure, cancer or any other condition that requires special treatment
* Relatives participating in the study
* Have plans to change residence
* Criteria of the researcher - for clinical reasons or adherence to the protocol
* Weight loss>5% of total body weight in the previous 4 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change in body weight | baseline to 3 months

SECONDARY OUTCOMES:
Change in body weight | baseline to 6 months
Change in body mass index | baseline to 3 months and baseline to 6 months
Change in waist circumference | baseline to 3 months and baseline to 6 months
Change in body fat percentage | baseline to 3 months and baseline to 6 months
Change in the Beck Depression Inventory Scale | baseline to 3 months and baseline to 6 months
  The Beck Depression Inventory (BDI) is a 21-item questionnaire that assesses mood over the previous week. Total scores range from 0 to 63, with higher values indicating more severe symptoms of depression. Scores of 0-9 reflect minimal (subclinical) symptoms, values of 10-18, 19-29, and ≥30 indicate mild, moderate, and severe symptoms of depression, respectively.
Change in the Short Form-36 Health Survey Score | baseline to 3 months and baseline to 6 months
  The SF-36 Health Survey evaluates aspects of quality of life in adult populations (over 16 years of age). The result of its application is the generation of eight concepts or scales of health, which is the result of the average of the sum of all questions contained in the questionnaire for each concept. These eight concepts are: physical function, physical role, corporal pain, general health, vitality, social function, emotional role and mental health. The SF-36 is a self-applied instrument and contains 36 questions. For each scale, the answer to each question is coded and recoded (10 questions), and the results are interpreted on a scale of 0 to 100, with lower scores indicating poorer health and higher scores better health.
Change in systolic and diastolic blood pressure | baseline to 3 months and baseline to 6 months
Change in fasting glucose | baseline to 3 months
Change in total cholesterol | baseline to 3 months
Change in LDL-cholesterol | baseline to 3 months
Change in HDL-cholesterol | baseline to 3 months
Change in triglycerides | baseline to 3 months
Change in gamma glutamyl transferase | baseline to 3 months
Number of participants achieving 5% of weight loss | baseline to 3 months and baseline to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de Promoción de Salud Nutricional (CPSN), Hermosillo, Sonora, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ruelas AL, Martinez Contreras TJ, Esparza Romero J, Diaz Zavala RG, Candia Plata MDC, Hingle M, Armenta Guirado B, Haby MM. Factors influencing adults to drop out of intensive lifestyle interventions for weight loss. Transl Behav Med. 2023 Apr 15;13(4):245-254. doi: 10.1093/tbm/ibac112. PMID 36694376